CLINICAL TRIAL: NCT03192826
Title: Study of the Efficacy of Brinzolamide 1% Plus Brimonidine 0.2% Versus Brimonidine 0.2% in the Prevention of Intraocular Pressure Rise After Nd-YAG Laser Capsulotomy
Brief Title: Brinzolamide/Brimonidine Combination vs Brimonidine 0.2% in the Prevention of IOP Rise After Nd-YAG Laser Capsulotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, MD, PhD, Associate Professor of Ophthalmology, Univerisity of Patras, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8393 / 26- 4- 2016
Record Dates: First submitted 2017-06-18; First posted 2017-06-20 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Posterior Capsule Opacification; Ocular Hypertension
Keywords: Nd-YAG capsulotomy; ocular hypertension; brimonidine; brinzolamide
MeSH Terms: conditions — Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double masked comparative study
Who Masked: Participant, Investigator
Masking Description: Patients are masked to their assignment by covering the labels on the bottles of the drugs administered The investigator responsible for the measurement of the intraocular pressure is also masked to the intervention administered to each patient.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Brinzolamide/Brimonidine FC (Active Comparator): 1 drop of Brinzolamide/Brimonidine FC 1 hour before capsulotomy
  Interventions: Drug: Brinzolamide/Brimonidine FC
- Brimonidine 0.2% (Active Comparator): 1 drop of Brimonidine 0.2% 1 hour before Nd-YAG capsulotomy
  Interventions: Drug: Brimonidine 0.2%
- Artificial tears (Placebo Comparator): 1 drop of artificial tears 1 hour before Nd-YAG capsulotomy
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Brinzolamide/Brimonidine FC — 1 drop of Brinzolamide/Brimonidine FC 1 hour before capsulotomy
  Other Names: SIMBRINZA (brinzolamide/brimonidine 1%/0.2%), Alcon Lab. Ltd
  Arms: Brinzolamide/Brimonidine FC
Drug: Brimonidine 0.2% — 1 drop of Brimonidine 0.2% 1 hour before Nd-YAG capsulotomy
  Other Names: ALPHAGAN (brimonidine tartrate 0.2%) Allergan Pharm. Ltd
  Arms: Brimonidine 0.2%
Drug: Artificial tears — 1 drop of artificial tears 1 hour before Nd-YAG capsulotomy
  Other Names: TEARS NATURALE EY.DRO.SOL 0.1%+0.3% Alcon Laboratories Ltd
  Arms: Artificial tears

SUMMARY:
To compare the efficacy of a Brinzolamide/Brimonidine fixed combination (FC) with Brimonidine 0.2% in preventing intraocular pressure (IOP) elevations after neodymium: yttrium-aluminum-garnet (Nd:YAG) laser posterior capsulotomy.

DETAILED DESCRIPTION:
In this prospective, randomized, double masked clinical trial, patients scheduled to undergo Nd:YAG laser posterior capsulotomy for posterior capsule opacification are randomized in 3 groups. The Brimonidine group receives 1 drop of Brimonidine 0.2%. The Brinzolamide/Brimonidine group receives 1 drop of Brinzolamide 1%/Brimonidine 0.2% fixed combination. The Control group receives artificial tears. All groups are administered a single drop instillation, approximately one hour before Nd:YAG application. Intraocular pressure measurements are performed before treatment (baseline) and at the 1, 3, 24 hours and 1 week post treatment.

Dexamethasone ophthalmic drops are prescribed q.i.d. for one week after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo laser posterior capsulotomy due to posterior capsule opacification (PCO) after uneventful phacoemulsification cataract extraction with implantation of posterior chamber intraocular lenses (IOL/PC).

Exclusion Criteria:

* baseline IOP greater than 21mmHg
* glaucomatous eyes, already under treatment with anti glaucomatic medications
* intraocular surgery except for uncomplicated cataract surgery
* previous photorefractive surgery
* active ocular inflammation or infection
* patients under systemic administration of medications known to affect IOP
* patients with severe respiratory or cardiovascular disease
* pregnant or breast feeding women, and individuals with known hypersensitivity or contraindication for administration of the medications tested
* a measurement of IOP > 30 mmHg at any time point of the study, or an increase from baseline >20 mmHg

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2017-07-08 (Actual); Study Completion 2017-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constantinos Georgakopoulos, MD, PhD, Study Director — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brinzolamide/Brimonidine FC | Brimonidine 0.2% | Artificial Tears
Started | 27 | 27 | 25
Completed | 27 | 27 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinzolamide/Brimonidine FC | Brimonidine 0.2% | Artificial Tears | Total
Number analyzed (Participants) | 27 | 27 | 25 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (6.3) | 65.2 (6.0) | 67.6 (3.9) | 65.5 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 13 | 37
  Male | 14 | 16 | 12 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 27 | 27 | 25 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 27 | 27 | 25 | 79

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) at 1 Hour After Nd-YAG Posterior Capsulotomy
Description: Comparison of intraocular pressure at 1 hour after Nd-YAG posterior capsulotomy compared to Baseline IOP
Time Frame: 1 hour
Population: Comparison of intraocular pressure at 1 hour after Nd-YAG posterior capsulotomy compared to Baseline IOP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brinzolamide/Brimonidine FC | Brimonidine 0.2% | Artificial Tears
Number analyzed (Participants) | 27 | 27 | 25
mmHg
  Baseline | 15.6 (1.5) | 15.7 (1.5) | 15.2 (1.9)
  1 hour | 13.7 (2.0) | 14.7 (3.7) | 19.5 (2.9)
Statistical Analysis 1: Comparison: Brinzolamide/Brimonidine FC vs Brimonidine 0.2% vs Artificial Tears; Test type: Equivalence — The SPSS statistical package version 23.0 (Statistical Package for the Social Sciences, version 23.0, SSPS Inc. Chicago, IL, USA) was used for statistical analysis; p < 0.05, ANOVA; Repeated measures ANOVA was used to compare parametric values with Bonferroni post hoc test for within group comparisons; Mean Difference (Final Values) = 0.05 — the reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance

2. Primary Outcome: Intraocular Pressure (IOP) at 3 Hours After Nd-YAG Posterior Capsulotomy
Description: Comparison of intraocular pressure at 3 hours after Nd-YAG posterior capsulotomy compared to Baseline IOP
Time Frame: 3 hours
Population: Comparison of intraocular pressure at 3 hours after Nd-YAG posterior capsulotomy compared to Baseline IOP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brinzolamide/Brimonidine FC | Brimonidine 0.2% | Artificial Tears
Number analyzed (Participants) | 27 | 27 | 25
mmHg
  Baseline | 15.6 (1.5) | 15.7 (1.5) | 15.2 (1.9)
  3 hours | 12.7 (1.5) | 14.7 (3.7) | 19.5 (2.9)
Statistical Analysis 1: Comparison: Brinzolamide/Brimonidine FC vs Brimonidine 0.2% vs Artificial Tears; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.05 — the reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance

3. Primary Outcome: Intraocular Pressure (IOP) at 24 Hourw After Nd-YAG Posterior Capsulotomy
Description: Comparison of intraocular pressure at 24 hours after Nd-YAG posterior capsulotomy compared to Baseline IOP
Time Frame: 24 hours
Population: Comparison of intraocular pressure at 24 hours after Nd-YAG posterior capsulotomy compared to Baseline IOP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brinzolamide/Brimonidine FC | Brimonidine 0.2% | Artificial Tears
Number analyzed (Participants) | 27 | 27 | 25
mmHg
  Baseline | 15.6 (1.5) | 15.7 (1.5) | 15.2 (1.9)
  24 hours | 14.6 (1.1) | 15.5 (1.7) | 15.8 (1.8)
Statistical Analysis 1: Comparison: Brinzolamide/Brimonidine FC vs Brimonidine 0.2% vs Artificial Tears; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.05 — the reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance

4. Primary Outcome: Intraocular Pressure (IOP) at 1 Week After Nd-YAG Posterior Capsulotomy
Description: Comparison of intraocular pressure at 1 week after Nd-YAG posterior capsulotomy compared to Baseline IOP
Time Frame: 1 week
Population: Comparison of intraocular pressure at 1 weekafter Nd-YAG posterior capsulotomy compared to Baseline IOP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brinzolamide/Brimonidine FC | Brimonidine 0.2% | Artificial Tears
Number analyzed (Participants) | 27 | 27 | 25
mmHg
  Baseline | 15.6 (1.5) | 15.7 (1.5) | 15.2 (1.9)
  1 week | 15.5 (1.1) | 15.3 (1.5) | 15.6 (1.7)
Statistical Analysis 1: Comparison: Brinzolamide/Brimonidine FC vs Brimonidine 0.2% vs Artificial Tears; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.05 — the reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance

ADVERSE EVENTS:
Time Frame: 1month
Description: The same with clinicaltrials.gov Definitions
Arm/Group | Brinzolamide/Brimonidine FC | Brimonidine 0.2% | Artificial Tears
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/25

LIMITATIONS AND CAVEATS:
Corneal thickness was not assessed. The measurement of IOP at more time points could have provided more information regarding the effect of BBFC. We could enroll a larger group of patients in order to provide more strength in our analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT03192826/Prot_SAP_000.pdf